CLINICAL TRIAL: NCT00014573
Title: Phase II Trial Of High Dose Cyclophosphamide, Cisplatin And Carmustine With Stem Cell Reconstitution Followed By Specific Cellular Therapy In Patients With Recurrent Or Refractory Brain Tumors
Brief Title: Chemotherapy and Vaccine Therapy Followed by Bone Marrow or Peripheral Stem Cell Transplantation and Interleukin-2 in Treating Patients With Recurrent or Refractory Brain Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068559; P30CA022453 (NIH); WSU-D-1654; WSU-07-92-98-P04-FB (Other: Wayne State University - Human Investigation Committee); NCI-G01-1937
Record Dates: First submitted 2001-04-10; First posted 2004-04-05 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood infratentorial ependymoma; childhood supratentorial ependymoma; childhood central nervous system germ cell tumor; recurrent adult brain tumor; adult brain stem glioma; adult medulloblastoma; adult glioblastoma; childhood high-grade cerebral astrocytoma; adult anaplastic astrocytoma; childhood choroid plexus tumor; childhood grade III meningioma; adult anaplastic ependymoma; adult mixed glioma; adult central nervous system germ cell tumor; adult ependymoblastoma; recurrent childhood brain stem glioma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; adult choroid plexus tumor; recurrent childhood ependymoma; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Medulloblastoma; Glioblastoma; Astrocytoma; Choroid Plexus Neoplasms; Ependymoma; Glioma; Neuroectodermal Tumors, Primitive; Familial ependymoma; Meningioma; Gliosarcoma | interventions — aldesleukin; FANG vaccine; Filgrastim; sargramostim; Carmustine; Cisplatin; Cyclophosphamide; Paclitaxel; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: aldesleukin
Biological: autologous tumor cell vaccine
Biological: filgrastim
Biological: sargramostim
Biological: therapeutic autologous lymphocytes
Drug: carmustine
Drug: cisplatin
Drug: cyclophosphamide
Drug: paclitaxel
Procedure: autologous bone marrow transplantation
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with bone marrow or peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells. Vaccines made from a person's white blood cells and tumor cells may make the body build an immune response to kill tumor cells. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and vaccine therapy followed by bone marrow or peripheral stem cell transplantation and interleukin-2 in treating patients who have recurrent or refractory brain cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effectiveness of induction paclitaxel and cyclophosphamide followed by autologous tumor cell vaccine and sargramostim (GM-CSF) followed by high-dose chemotherapy with cisplatin, cyclophosphamide, and carmustine, autologous bone marrow or peripheral blood stem cell transplantation, and interleukin-2 in patients with recurrent or refractory primary high-grade brain tumors.
* Determine the safety and toxicity of this regimen in these patients.
* Determine if a specific quantitative cellular response can be elicited in patients treated with this regimen.

OUTLINE: After partial surgical resection of tumor, patients receive induction chemotherapy comprising paclitaxel IV over 3 hours and cyclophosphamide IV over 1 hour on day 1. Patients also receive filgrastim (G-CSF) subcutaneously (SC) daily beginning on day 3 and continuing until peripheral blood stem cell (PBSC) or bone marrow collection is completed.

After the collection of PBSC or bone marrow, patients receive autologous tumor cell vaccine and sargramostim (GM-CSF) SC once every 2 weeks for up to 5 vaccinations. Two weeks after the last vaccination, patients undergo a second leukapheresis to collect lymphocytes.

After completion of the second leukapheresis, patients receive high-dose chemotherapy comprising cisplatin IV continuously over 24 hours on day -5, cyclophosphamide IV over 1 hour on days -5, -4, and -3, and carmustine IV over 2 hours on day -2. Patients undergo autologous bone marrow or PBSC transplantation on day 0. Patients receive G-CSF IV daily beginning on day 0 and continuing until blood counts recover.

Approximately 12 weeks after bone marrow or PBSC transplantation, patients receive autologous lymphocytes IV over 2-5 hours. Patients also receive interleukin-2 IV once every other day for 10 days.

Patients are followed at 18, 24, 36, 40, and 52 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed active recurrent or refractory primary high-grade brain tumor

  * Tumor must be surgically accessible
* Bidimensionally measurable disease by clinical exam, CT scan, or x-ray

  * Disease must be outside a previously irradiated field or have progressed or developed after radiotherapy
  * Previously treated metastatic bony lesions are not considered measurable
  * No previously irradiated metastatic disease site unless no response or clear progression on imaging

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* CALGB 0-2

Life expectancy:

* More than 3 months

Hematopoietic:

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Liver function less than 2.5 times normal unless due to disease
* No active hepatitis B or C

Renal:

* Creatinine less than 1.5 mg/dL
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Left ventricular ejection fraction greater than 50% by MUGA or 2-D echocardiogram
* Electrocardiogram normal

Pulmonary:

* FEV1 and DLCO greater than 50% predicted OR
* Clearance by pulmonologist

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No serious underlying co-morbid disease or other medical or psychiatric factor that would preclude study
* Able to be weaned off steroids after surgery

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Recovered from prior conventional chemotherapy

Endocrine therapy:

* No concurrent steroid therapy for mass effect

Radiotherapy:

* See Disease Characteristics
* Recovered from prior conventional radiotherapy

Surgery:

* See Disease Characteristics

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-08; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Abella, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States